CLINICAL TRIAL: NCT03778411
Title: Non-invasive Evaluation of Portal Hypertension in Patients With Compensated Advanced Chronic Liver Disease by Assessment of Spleen Stiffness Using Vibration Controlled Transient Elastography
Brief Title: Non-invasive Evaluation of Portal Hypertension in Patients With Compensated Advanced Chronic Liver Disease by Assessment of Spleen Stiffness Using VCTE by FibroScan.
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Echosens (Industry)
Responsible Party: Principal Investigator, Raj Vuppalanchi, Associate Professor of Medicine, Indiana University
Other Study IDs: 1804223843
Record Dates: First submitted 2018-08-30; First posted 2018-12-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Chronic Liver Disease, NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- cACLD: 200 people with compensated advanced chronic liver disease who have not undergone liver transplant
  Interventions: Device: VCTE with splenic stiffness measurement
- cACLD-post transplant: 100 people with compensated advanced chronic liver disease who have previously undergone liver transplant
  Interventions: Device: VCTE with splenic stiffness measurement

INTERVENTIONS:
Device: VCTE with splenic stiffness measurement — Subjects will undergo vibration controlled transient elastography to measure liver stiffness (LSM) liver steatosis via controlled attenuation parameter (CAP) and splenic stiffness

SUMMARY:
Hypothesis: The severity of portal hypertension in compensated advanced chronic liver disease (cACLD) can be assessed using vibration controlled transient elastography (VCTE) via the FibroScan® 502 Touch by measuring SS (splenic stiffness) Specific Aims: SS by VCTE will be measured in this single center clinical study comprising of 200 patients with cACLD (deﬁned by LSM ≥10 kilopascals (kPa) according to the Baveno VI recommendations) who have not had a liver transplant and 100 subjects who are post-liver transplant. The association between baseline SS values will be examined in relation to the manifestations of portal hypertension such as esophageal or gastric varices.

Specific Aim: To examine the relationship between SS and the presence of esophageal and gastric varices in patients with compensated advanced chronic liver disease (cACLD).

Proposed Study Design: This is a cross sectional study that evaluates the relationship between SS by VCTE in patients with cACLD and manifestations of portal hypertension.

DETAILED DESCRIPTION:
A new term, compensated advanced chronic liver disease (cACLD) defining patients in the early phases of severe chronic liver disease, including both patients with severe fibrosis or pre-cirrhotic patients and patients with compensated cirrhosis is considered very helpful for both clinical practice and research purposes. Cirrhosis should no longer be regarded as a terminal disease and the concept of a dynamic process is increasingly accepted.

Currently, the management of patients with cACLD includes assessment for severity of portal hypertension and risk stratification. Cirrhosis is currently classiﬁed into two main prognostic stages: compensated and decompensated cirrhosis. This classiﬁcation depends on the presence or absence of clinically evident decompensating events (speciﬁcally ascites, variceal hemorrhage, and encephalopathy). The Child-Turcotte-Pugh (CTP) classiﬁcation has been used to stratify patients with cirrhosis. Patients with cirrhosis belonging to the CTP-A class are compensated, whereas those in the CTP-B/C class are mostly decompensated. Similarly, Model for End-Stage Liver Disease (MELD) is a reliable measure of mortality risk in patients with end-stage liver disease and used to help prioritize organ allocation for transplant. However, MELD scores of <10, typically seen in CTP-A, are unlikely to have prognostic value as the likelihood of clinical events in a 1 to 2-year time frame is low. Therefore, both CTP and MELD scores best stratify cirrhosis patients with decompensation and have limited use in compensated cirrhotics who have no liver-related symptoms.

Patients with compensated cirrhosis are sub-staged based on the severity of portal hypertension. However, measurement of portal pressure through direct puncture of the portal vein is risky and not routinely performed. Therefore, portal pressure is assessed indirectly by calculation of hepatic vein pressure gradient (HVPG) by measuring the difference between wedge and free hepatic venous pressure.The normal value of HVPG is between 3 and 5 mmHg. Currently, the severity of portal hypertension is defined as mild when HVPG is 6 but <10 mm Hg, ≥10 mm Hg as clinically significant portal hypertension (CSPH), and ≥12 mm Hg as severe portal hypertension (SPH). Evaluation of a compensated cirrhotic by HVPG is ideal for risk stratification as CSPH is associated with an increased risk of varices, decompensation (ascites, variceal hemorrhage and/or hepatic encephalopathy) and hepatocellular cancer. However, measurement of HVPG is cumbersome, invasive, non-standardized and often limited to tertiary care centers due to limited expertise. Therefore, there is a need for non-invasive tools that can estimate HVPG easily, reproducibility and with high diagnostic accuracy.

Liver stiffness measurement (LSM) by vibration controlled transient elastography (VCTE) is currently used for non-invasive diagnosis liver fibrosis in patients with NAFLD (non alcoholic fatty liver) and NASH (non alcoholic steatohepatitis). In patients with cirrhosis, LSM is likely indicative of cumulative stiffness from underlying liver fibrosis and portal hypertension. Portal hypertension-related splenomegaly is frequently accompanied by patients with cirrhosis due to portal venous congestion and hyperplasia of splenic tissue, and its usefulness for diagnosis of portal hypertension has been studied. However, the direct relationship between the size of the spleen and the severity of portal hypertension is still under debate. Recent studies have focused on ultrasound-based measurement of spleen stiffness (SS) as it is reflective of portal hypertension-related changes in the spleen, including splenomegaly. Measurement of SS has also accurately predicted both the presence of varices and the degree of portal hypertension. Spleen Stiffness (SS) by VCTE is an emerging tool for assessment of portal hypertension and its feasibility has been reported both in adults and children.

FibroScan is a diagnostic device based on VCTE. It measures a mean tissue stiffness (between 25 mm and 65 mm in the liver of non-obese patients) in a medium considered as homogeneous and isotropic. FibroScan is equipped with a probe composed of an ultrasonic transducer (3.5 MHz for non-obese patients) mounted on the axis of a vibrator. This vibrator generates a low-frequency pulse (50 Hz and 2 mm peak-to-peak amplitude for LS measurement in non-obese patients) that induces a shear wave that propagates through the tissue. Shear wave propagation is followed by pulse-echo ultrasound and the strains induced in the tissue are computed as a function of time and depth. Tissue stiffness E is deduced from the shear wave speed (SWS or Vs) obtained by measuring the slope of the shear wave on the strain matrix using a time-of-flight algorithm (E = 3ρVs² where ρ is the body mass of the tissue). In soft tissues, the body mass is close to the one of water. A body mass ρ of 1,000 kg/m3 was used for the density of the spleen. The ultrasound acquisition is performed between 20 mm and 80 mm below skin surface and the measurement is performed between 25 mm and 55 mm. The stiffness of the spleen ranges between 5 kPa and 100 kPa. It is currently undergoing regulatory approval as a diagnostic tool for non-invasive assessment of portal hypertension.

The natural history of NASH or other chronic liver disorders with advanced fibrosis/ cirrhosis across the different clinical stages of cirrhosis is currently not well understood. Therefore, non-invasive tools that can assess the severity of cirrhosis and risk stratify prior to decompensation is currently an unmet need. Simultaneous assessment of LSM and SS using VCTE may eventually allow for a noninvasive, immediate, objective and efficient method for estimation of disease severity in patients with NASH cirrhosis. Moreover, assessment over time of LSM and SS may also allow for assessment of disease progression or regression from treatment interventions. It is anticipated that baseline measurements of SS/LSM and longitudinal changes (ΔSS/Δt or ΔLSM/Δt) will serve as a prognostic tool in patients with cACLD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Ability to provide informed consent
3. Previous Fibroscan with LSM ≥10 kilopascals (kPa)

Exclusion Criteria:

1. Inability or refusal to provide informed consent
2. Fasting for less than three hours prior to the scan
3. Subject is a pregnant or lactating female
4. Subject with current, significant alcohol consumption
5. Subject is unable to reliably quantify alcohol consumption based upon local study physician judgment
6. Patients with a pacemaker or defibrillator
7. Acute hepatitis defined as AST/ALT > 500 U/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with compensated advanced chronic liver disease (deﬁned by LSM ≥10 kilopascals (kPa) who have not had a liver transplant and 100 subjects with compensated advanced chronic liver disease who are post-liver transplant.
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Risks of decompensation | Two years
  The relationship between splenic stiffness (SS) and the presence of esophageal and gastric varices in patients with compensated advanced chronic liver disease (cACLD) will be measured with VCTE by the CAP score.
  CAP is measured in dB/M, with a score range from 100-400. A score of 225 or less is considered to indicate a normal amount of fat in the liver. As the score increases, the amount of steatosis (fat) in the liver is also thought to be elevated.

SECONDARY OUTCOMES:
Risks of decomposition | Two years
  The relationship between splenic stiffness (SS) and the presence of esophageal and gastric varices in patients with compensated advanced chronic liver disease (cACLD) will be measured with VCTE with splenic stiffness score.
  VCTE is measured in units of kPA with a score range from 0-75. An increased number is generally associated with a higher level of liver scarring, but the ranges are based on the underlying liver disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No